CLINICAL TRIAL: NCT03927118
Title: The Effect of Dexamethasone Implant on Retinal Nerve Fiber and Optic Disc Morphology in Patients With Diabetic Maculopathy
Brief Title: Effect of Dexamethasone Implant on Optic Disc
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Atilla Alpay, Associate professor, Bulent Ecevit University
Other Study IDs: BulentEU2
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Glaucoma and Ocular Hypertension; Diabetic Macular Edema; Intravenous Drug Usage; Optic Disk Disorders
Keywords: Diabetic maculopathy; dexamethasone implant; optic disc; vascular endothelial growth factor
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: intravitreal dexamethasone implant application — Peripapillary RNFL thickness measurements and colored fundus photographs were compared before and 6 months after intravitreal DEX implant injection. The cup-to-disc ratios of fundus photographs were calculated using the Image-J program.
  Other Names: The Effect of Dexamethasone Implant on Retinal Nerve Fiber and Optic Disc in Diabetic maculopathy.

SUMMARY:
This study evaluates the effect of dexamethasone implant which is an intraocular corticosteroid on the optic nerve fibers. Retinal nerve fiber thicknesses and optic nerve head pitting rates were measured before and 6 months after the injection.

DETAILED DESCRIPTION:
Diabetic macular edema is the most frequent ocular complication of diabetes resulting in irreversible loss of vision if untreated. Dexamethasone implant implant is used to treat macular edema due to diabetes. It stay in the vitreous for 6 months after intravitreal administration.

Dexamethasone implant can lead to retinal nerve fiber layer and optic nerve damage by both increasing intraocular pressure and its direct effect on neural tissue during the effective 6-month period.

ELIGIBILITY:
Inclusion Criteria

Patients who underwent first time intravitreal injection

Exclusion Criteria

Previously received any surgery

Proliferative diabetic retinopathy

Glaucoma or glaucoma suspicion

Optic disc fatigue

Optic disc edema

Uveitis and media opacity

Blurred of image clarity

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals over 20 years of age were included in the study.
Study Population: Diabetic patient group will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Peripapillary RNFL thickness measurements | six month
  micrometer

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Alpay, Ass. Prf., Study Director — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bülent Ecevit Üniversitesi., Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du JH, Li X, Li R, Xu L, Ma RR, Liu SF, Zhang Z, Sun HZ. Elevation of serum apelin-13 associated with proliferative diabetic retinopathy in type 2 diabetic patients. Int J Ophthalmol. 2014 Dec 18;7(6):968-73. doi: 10.3980/j.issn.2222-3959.2014.06.10. eCollection 2014. PMID 25540748
- [Background] Liu L, Wu X, Liu L, Geng J, Yuan Z, Shan Z, Chen L. Prevalence of diabetic retinopathy in mainland China: a meta-analysis. PLoS One. 2012;7(9):e45264. doi: 10.1371/journal.pone.0045264. Epub 2012 Sep 20. PMID 23028893
- [Background] Assmann TS, Brondani LA, Boucas AP, Rheinheimer J, de Souza BM, Canani LH, Bauer AC, Crispim D. Nitric oxide levels in patients with diabetes mellitus: A systematic review and meta-analysis. Nitric Oxide. 2016 Dec 30;61:1-9. doi: 10.1016/j.niox.2016.09.009. Epub 2016 Sep 24. PMID 27677584
- [Background] Suwanpradid J, Rojas M, Behzadian MA, Caldwell RW, Caldwell RB. Arginase 2 deficiency prevents oxidative stress and limits hyperoxia-induced retinal vascular degeneration. PLoS One. 2014 Nov 6;9(11):e110604. doi: 10.1371/journal.pone.0110604. eCollection 2014. PMID 25375125
- [Background] Celik M, Cerrah S, Arabul M, Akalin A. Relation of asymmetric dimethylarginine levels to macrovascular disease and inflammation markers in type 2 diabetic patients. J Diabetes Res. 2014;2014:139215. doi: 10.1155/2014/139215. Epub 2014 Apr 3. PMID 24804267
- [Background] Lluch P, Segarra G, Medina P. Asymmetric dimethylarginine as a mediator of vascular dysfunction in cirrhosis. World J Gastroenterol. 2015 Aug 28;21(32):9466-75. doi: 10.3748/wjg.v21.i32.9466. PMID 26327755
- [Background] Heunisch F, Chaykovska L, von Einem G, Alter M, Dschietzig T, Kretschmer A, Kellner KH, Hocher B. ADMA predicts major adverse renal events in patients with mild renal impairment and/or diabetes mellitus undergoing coronary angiography. Medicine (Baltimore). 2017 Feb;96(6):e6065. doi: 10.1097/MD.0000000000006065. PMID 28178159
- [Background] Franceschelli S, Ferrone A, Pesce M, Riccioni G, Speranza L. Biological functional relevance of asymmetric dimethylarginine (ADMA) in cardiovascular disease. Int J Mol Sci. 2013 Dec 16;14(12):24412-21. doi: 10.3390/ijms141224412. PMID 24351825
- [Background] Yin YL, Zhu ML, Wan J, Zhang C, Pan GP, Lu JX, Ping S, Chen Y, Zhao FR, Yu HY, Guo T, Jian X, Liu LY, Zhang JN, Wan GR, Wang SX, Li P. Traditional Chinese medicine xin-mai-jia recouples endothelial nitric oxide synthase to prevent atherosclerosis in vivo. Sci Rep. 2017 Mar 2;7:43508. doi: 10.1038/srep43508. PMID 28252100
- [Background] Marcovecchio ML, Widmer B, Turner C, Dunger DB, Dalton RN. Asymmetric dimethylarginine in young people with Type 1 diabetes: a paradoxical association with HbA(1c). Diabet Med. 2011 Jun;28(6):685-91. doi: 10.1111/j.1464-5491.2011.03252.x. PMID 21294768
- [Background] Ersoy B, Eroglu N, Cetin M, Onur E, Ozkol M, Coskun S. Asymmetric dimethylarginine levels and diabetes duration: Relationship with measures of subclinical atherosclerosis and cardiac function in children and adolescents with Type 1 diabetes. Diab Vasc Dis Res. 2018 May;15(3):196-203. doi: 10.1177/1479164118757921. Epub 2018 Mar 2. PMID 29498294
- [Background] Lin KY, Ito A, Asagami T, Tsao PS, Adimoolam S, Kimoto M, Tsuji H, Reaven GM, Cooke JP. Impaired nitric oxide synthase pathway in diabetes mellitus: role of asymmetric dimethylarginine and dimethylarginine dimethylaminohydrolase. Circulation. 2002 Aug 20;106(8):987-92. doi: 10.1161/01.cir.0000027109.14149.67. PMID 12186805